CLINICAL TRIAL: NCT02999139
Title: Analytic, Prospective Cohort Study of Athletes Enrolled in an Exercise Training Intervention
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Daisuke Sugimoto, Lead Research Technologist, Boston Children's Hospital
Other Study IDs: P00023758
Record Dates: First submitted 2016-12-14; First posted 2016-12-21 (Estimated); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Exercise Training
Keywords: Injury; Prevention
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- ACL Return to Play: A specific training program, with emphasis on hamstring strengthening. There will also be a specificity on pivoting and jumping safely.
- Gait Retraining: Will receive training that is specific to running. Drills will help enforce a more efficient running form, as well as strengthening important muscle groups such as the hip abductors and adductors.
- Private Training: Participants will receive a broad training program, targeting all major muscle groups. The goal is to increase muscle strength, mobility and aerobic capacity to reduce the risk of injury.

SUMMARY:
Participants who train at The Micheli Center for Sports Injury Prevention, will undergo testing of muscular strength, range of motion, flexibility, aerobic capacity and muscular endurance. They will complete training with a certified trainer and injury prevention specialist until their specific goals are meet. Upon completion of training, they will fill out an injury questionnaire every three months for five to ten years.

ELIGIBILITY:
Inclusion Criteria:

* Males, Females, age 6 and over

Exclusion Criteria:

* younger than 6 years old

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Male and females age 6 and over.
Sampling Method: Probability Sample
Enrollment: 633 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-29 (Actual)

PRIMARY OUTCOMES:
Injury | After a subject undergoes training at The Micheli Center for Sports Injury Prevention, they will complete a survey every 3 months for the next 10 years.
  For purposes of our study, an injury is one that:
  1. occurred as a result of participation in sport AND
  2. required medical attention by a team athletic trainer or a physician AND
  3. resulted in restriction of the student-athlete's participation for one or more days beyond the day of injury OR
  4. resulted in any fracture, concussion, or dental injury regardless of whether or not it resulted in restriction of the student-athlete's participation

SECONDARY OUTCOMES:
Training Habits | After a subject undergoes training at The Micheli Center for Sports Injury Prevention, they will complete a survey every 3 months for the next 10 years.
  Surveys will answer if participants continue with their new training habits
Muscular Strength | Before training and after completion of training at The Micheli Center for Sports Injury Prevention. Training can last from four weeks to a year.
  This will be measured by hand held dynamometer pre and post training intervention. Will testing major muscles such as the quadriceps, hamstrings, biceps, triceps.
Aerobic Capacity | Before training and after completion of training at The Micheli Center for Sports Injury Prevention. Training can last from four weeks to a year.
  This will be estimated by the step test, done pre and post training.
Anaerobic Capacity | Before training and after completion of training at The Micheli Center for Sports Injury Prevention. Training can last from four weeks to a year.
  This will be measured by a series of tests such as the vertical jump test and shuttle run. These measures will be tested pre and post training.
Range of Motion | Before training and after completion of training at The Micheli Center for Sports Injury Prevention. Training can last from four weeks to a year.
  This will be measured by goniometer at different joints such as the knee and ankle pre and post training.

CONTACTS AND LOCATIONS:
Locations (1):
- The Micheli Center for Sports Injury Prevention, Waltham, Massachusetts, United States